CLINICAL TRIAL: NCT04773795
Title: Evaluation of EndoZip System in Obese Patients Who Failed to Reduce Weight With Non-surgical Weight-loss Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitinotes Surgical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL00003
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoZip System (Experimental): The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (4-8) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.
  Interventions: Device: EndoZip System

INTERVENTIONS:
Device: EndoZip System — The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (4-8) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.

SUMMARY:
A multicenter, prospective, single-arm, open-label, controlled clinical trial aimed to evaluate the safety and effectiveness of the EndoZip system procedure, coupled with lifestyle modifications, for weight reduction in obese patients with BMI of 30-40 kg/m2.

DETAILED DESCRIPTION:
study will include up to 45 (10-20 patients per site), ages of 21 -70 of obese patients who failed to reduce weight with non-surgical weight-loss methods.

The duration for each participant will be 12 months and will include the following follow up visits and procedures:

* Office visits: screening, 1 week, and 1, 2, 4, 6, 8, 10, and 12 month(s)
* Remote follow up (by Phone): 3, 5, 7, 9, and 11 month(s)
* Endoscopy procedure: baseline, 2 and 6 months post EndoZip procedure
* Motility evaluation by Gastric Emptying Breath Test (GEBT): baseline, 6 months
* Physical examination, vital signs, waist circumference and BMI: baseline, 1 week, 1, 2, 4, 6, 8, 10 and 12 months
* Blood tests: baseline,2, 6 and 12 months
* IWQOL-Lite: baseline, 2, 6 and 12 months
* Psychological health questionnaire-9 (PHQ-9) :baseline
* Sleep Apnea (only for the relevant population): baseline 2, 6 and 12 months

The patient will required to follow a specific diet and to have a physical activity during the study period ( 12 month).

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70
2. BMI ≥ 30 and ≤40 kg/m².
3. Willingness to comply with the substantial behavioral modifications program as required by the procedure.
4. Patients with history of failure with non-surgical weight-loss methods.
5. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, completing IWQOL questionnaire and completing the medically supervised diet and behavior modification program.
6. Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow- up visits.
7. Ability to give informed consent.
8. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.

Exclusion Criteria:

1. Prior surgery of any kind on the gastrointestinal tract (except uncomplicated cholecystectomy or appendectomy).
2. Patients with history of small bowel or colonic obstruction, and/or adhesive peritonitis and/or abdominal adhesions.
3. Patients with any inflammatory disease
4. Patients with history of cancer in the gastrointestinal tract.
5. Potential upper gastrointestinal bleeding conditions such as a history of angioectasias.
6. A known gastric mass or gastric polyps > 1 cm in size.
7. Patients with TG >500 or LDL >190
8. A known hiatal hernia > 4cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms while on maximal medical therapy.
9. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope.
10. Patient with motility disorders of the GI tract or intractable constipation
11. Patients with known coagulation disorder (INR >1.5) or on anticoagulation therapy.
12. Type 1 diabetes or Type 2 diabetes with a HgbA1c >8 in 6 weeks prior the procedure or use of any medication for diabetes other than metformin. Patients with any serious health condition unrelated to their weight that would increase the risk of endoscopy
13. Patients with chronic abdominal pain
14. Patients with hepatic insufficiency or cirrhosis
15. Patients that used an intragastric device for weight loss within 2 years prior to this study.
16. Patients with psychological health questionnaire-9 (PHQ-9) score of 10 or higher.
17. Patients receiving daily prescribed treatment with high dose aspirin (> 100mg daily), anti-inflammatory agents, anticoagulants or other gastric irritants.
18. Patients with history or current abuse of drugs or alcohol
19. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication
20. egg, milk, or wheat allergy (unable to go through the GEBT)
21. Patients who are pregnant or breast-feeding.
22. Patients who are taking medications that cause weight loss
23. Patients with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 12 months, poorly-controlled hypertension, required use of NSAIDs
24. Patients taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications
25. Patients who are taking corticosteroids, immunosuppressants, and narcotics
26. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
27. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (severe COPD), pneumonia or cancer.
28. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, HIV, erythematous, scleroderma) or immunocompromised.
29. Specific diagnosed genetic disorder such as Prader Willi syndrome (motility disorder)
30. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating
31. Known history of endocrine disorders affecting weight such as uncontrolled hypothyroidism.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Peled, Study Director — NiTiNotes Ltd
Locations (1):
- Hospital Universitario HM Sanchinarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boskoski I, Lopez-Nava G, Ravishankar A, Bove V, Matteo MV, De Siena M, Pontecorvi V, Giannetti G, Iaconelli A, Spada C, Shamah SE. Automatic endoscopic gastroplasty for the treatment of obesity: results from a prospective multicenter study (with video). Gastrointest Endosc. 2025 Apr;101(4):818-827. doi: 10.1016/j.gie.2024.09.026. Epub 2024 Sep 21. PMID 39307402

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoZip System: The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (4-8) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.
  EndoZip System: The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (4-8) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.
Period: Overall Study
Arm/Group | EndoZip System
Started | 48
Completed | 45
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: patients undergo EndoZip procedure
Arm/Group | EndoZip System
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.13 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Total Body Weight Loss (kg) From Baseline to12 Months
Description: Change in body total body weight loss (kg) from baseline to 12 months post EndoZip procedure
Time Frame: 12 month
Measure: Mean (Standard Error); unit: kg
Arm/Group | EndoZip System
Number analyzed (Participants) | 45
kg | 13.2 (1.5)

2. Primary Outcome: Percentage of Patients With a Reduction in %TBWL of at Least 5% From Baseline to 12 Months.
Description: Percentage of patients with a reduction in %TBWL of at least 5% from baseline to 12 months.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | EndoZip System
Number analyzed (Participants) | 45
Participants | 34

ADVERSE EVENTS:
Time Frame: 1 year after the EndoZip procedure
Arm/Group | EndoZip System
All-Cause Mortality (participants affected / at risk) | 3/45
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 2/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoZip System (N=45)
Bleeding next to the suture area (Surgical and medical procedures) | 1 (1) — at suture number 4 a technical failure of insufficient proximal clip closer, led to an active bleeding, closed by endoscopic placement of 4 clips. The event was resolved within 72 hours with no clinical sequelae.
Mild Gastric perforation (Surgical and medical procedures) | 1 (1) — due to human error the physician didn't pull wire A to release the corset wire prior to system retrieval, as a result of the force exerted by the physician a part of the Bougie broke, also a gastric perforation was suspected
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoZip System (N=45)
abdominal pain (Surgical and medical procedures) | 1 (1)
anemic (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT04773795/Prot_SAP_000.pdf